CLINICAL TRIAL: NCT00929539
Title: A Phase II, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy, Safety and Tolerability of JTT-130 in Treatment-naïve, Metformin Only or Metformin Plus Sulfonylurea-treated Obese Type 2 Diabetic Patients
Brief Title: Safety and Efficacy Study of JTT-130 in Obese Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akros Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AT130-G-08-006
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Type II Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — diethyl 2-((3-dimethylcarbamoyl-4-((4'-trifluoromethylbiphenyl-2-carbonyl)amino)phenyl)acetyloxymethyl)-2-phenylmalonate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose 1 JTT-130 (Experimental)
  Interventions: Drug: JTT-130
- Dose 2 JTT-130 (Experimental)
  Interventions: Drug: JTT-130
- Dose 3 JTT-130 (Experimental)
  Interventions: Drug: JTT-130
- Placebo (Placebo Comparator)
  Interventions: Drug: JTT-130 Placebo

INTERVENTIONS:
Drug: JTT-130 — Tablets
  Arms: Dose 1 JTT-130; Dose 2 JTT-130; Dose 3 JTT-130
Drug: JTT-130 Placebo — Tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of JTT-130 on diabetes as well as the safety and tolerability of JTT-130 in obese Type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Have type 2 diabetes;
2. Body mass index (BMI) of > 27.0 kg/m2 and ≤ 45.0 kg/m2;
3. Are either drug naïve with respect to hypoglycemic agents OR are currently being treated with metformin alone or in combination with a sulfonylurea. Metformin and sulfonylurea dosing must be stable.

Exclusion Criteria:

1. Females who are pregnant or breast-feeding
2. Known medical history or presence of type 1 diabetes, pancreatitis, unstable or rapidly progressing retinopathy, nephropathy or neuropathy;
3. Acute coronary syndrome or uncontrolled hypertension;
4. Does not meet medication restriction criteria, as described in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2009-06; Primary Completion 2010-05 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in glycosylated hemoglobin (HbA1c) levels | End of Study

SECONDARY OUTCOMES:
Safety and tolerability data | End of Study

CONTACTS AND LOCATIONS:
Locations (62):
- United States (48):
  - Birmingham, Alabama
  - Muscle Shoals, Alabama
  - Scottsboro, Alabama
  - Tucson, Arizona
  - Encino, California
  - Los Angeles, California
  - Sacramento, California
  - Spring Valley, California
  - Valley Village, California
  - Walnut Creek, California
  - Waterbury, Connecticut
  - Delray Beach, Florida
  - Hialeah, Florida
  - Miami, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Sandy Springs, Georgia
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Erlanger, Kentucky
  - Lexington, Kentucky
  - Louisville, Kentucky
  - Madisonville, Kentucky
  - Paducah, Kentucky
  - New Hyde Park, New York
  - Greensboro, North Carolina
  - Morehead City, North Carolina
  - Statesville, North Carolina
  - Cincinnati, Ohio
  - Marion, Ohio
  - Tulsa, Oklahoma
  - Eugene, Oregon
  - Portland, Oregon
  - Charleston, South Carolina
  - Greer, South Carolina
  - North Charleston, South Carolina
  - Bristol, Tennessee
  - Austin, Texas
  - Corpus Christi, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Manassas, Virginia
  - Richmond, Virginia
  - Bellevue, Washington
  - Olympia, Washington
  - Oregon, Wisconsin
- Czechia (6):
  - Beroun
  - Brno
  - Ostrava
  - Pardubice
  - Prague
  - Velké Hoštice
- Hungary (2):
  - Sátoraljaújhely
  - Szikszó
- Netherlands (2):
  - Eindhoven
  - Groningen
- Russia (4):
  - Arkhangelsk
  - Moscow
  - Nizhny Novgorod
  - Saint Petersburg